CLINICAL TRIAL: NCT03117400
Title: Visible Vessels do Not Predict Clinically Significant Bleeding After EMR - a Systematic Description of the Post EMR Defect
Brief Title: Systematic Description of the Post EMR Defect
Status: Completed | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Clinical Professor, Western Sydney Local Health District
Other Study IDs: HREC/15/5/5.3 (4272)
Record Dates: First submitted 2017-04-11; First posted 2017-04-18 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Delayed Bleeding Post EMR; Large Laterally Spreading Lesion in the Colon; Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bland blue defect: The defect after endoscopic mucosal resection of the colonic large laterally spreading lesion (20mm or more) is blue without any other defect features (as described in the second group, 'non bland blue defect'). The blue is the result of the submucosal injection of dye (indigo carmine), used to lift lesions before starting the resection.
- Non bland blue defect: The defect after endoscopic mucosal resection of the colonic large laterally spreading lesion (20mm or more) is not just blue, but contains other defect features, such as visible vessels, herniation of vessels, submucosal fat, exposed muscle, fibrous bands, submucosal haemorrhage or non stained submucosa.

SUMMARY:
To date there are no available data on the utility of the endoscopic mucosal resection (EMR) defect in stratifying the risk of immediate or delayed adverse outcomes, particularly clinically significant post EMR bleeding (CSPEB).

The investigators aimed to analyse the data to determine if any of these EMR defect features allow us to estimate the risk of CSPEB. This will help endoscopists to identify defects with a high risk of adverse outcomes and may translate into improved patient outcomes.

DETAILED DESCRIPTION:
CSPEB is the most frequent serious complication after wide-field EMR of laterally spreading lesions ≥ 20mm (LSLs). There is no proven therapy for CSPEB and it remains a significant drawback of EMR. Visible vessels within the post EMR defect (PED) present themselves as logical targets for prophylactic treatment to prevent CSPEB. However, the clinical significance of these vessels is largely unknown. In the majority of studies risk factors identified for CSPEB include right colon location, lesion size and aspirin use. The investigators aimed to systematically describe and evaluate the clinical significance of the various endoscopic features of the post EMR defect PED including visible vessels.

A prospective study of LSLs ≥ 20mm referred for EMR at a single tertiary referral center will be performed.

Data collection includes patient, procedural and lesion characteristics. In all cases a systematic description of the PED is undertaken. The data of particular interest to this study includes: use of blood thinners, PED features including size, number and herniation of visible vessels, submucosal haemorrhage, fibrosis, fat and exposed muscle and the rate of CSPEB.These features were analysed for significant association with CSPEB. CSPEB was defined as any bleeding occurring after the completion of the procedure necessitating emergency department presentation, hospitalization or reintervention. CSPEB was compared to features of the PED to detect significant associations, using chi2 or Fisher's exact tests. Significant univariate variables will be taken forward for binomial logistic regression modelling.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for EMR of a LSL 20mm or larger
* Signed the informed consent

Exclusion Criteria:

* Clips used during the EMR procedure to close the defect, totally or partially
* Inadequate images to adequately assess the defect
* Use of blood thinners which have not been ceased according to the current guidelines for EMR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with a colonic laterally spreading lesion ≥ 20mm referred for EMR at a single tertiary referral centre will be included.
Sampling Method: Non-Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2013-05-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Defect features predicting clinically significant post EMR bleeding | day of procedure until 2 weeks after the procedure
  To assess if any of the defect features can predict clinically significant post EMR bleeding

SECONDARY OUTCOMES:
Defect features predicting other adverse events | day of procedure until 2 weeks after the procedure
  To assess if any of the defect features can predict perforation or recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, MBBS, FRACP, Principal Investigator — WSLHD
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desomer L, Tate DJ, Bahin FF, Awadie H, Chiang B, Holt B, Byth K, Bourke MJ. A systematic description of the post-EMR defect to identify risk factors for clinically significant post-EMR bleeding in the colon. Gastrointest Endosc. 2019 Mar;89(3):614-624. doi: 10.1016/j.gie.2018.11.023. Epub 2018 Nov 29. PMID 30503846